CLINICAL TRIAL: NCT03906630
Title: Comparison of the Accuracy of Telehealth Examination Versus Clinical Examination in the Detection of Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00101866
Record Dates: First submitted 2019-04-05; First posted 2019-04-08 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shoulder patients
  Interventions: Diagnostic Test: Telehealth clinical exam; Diagnostic Test: Standard clinical exam

INTERVENTIONS:
Diagnostic Test: Telehealth clinical exam — This is a pseudo telehealth clinical exam for patients presenting with shoulder pain
Diagnostic Test: Standard clinical exam — This is a standard in-person clinical exam for patients presenting with shoulder pain

SUMMARY:
The purpose of this study is to compare how accurately a pseudo-telehealth shoulder examination diagnoses rotator cuff tears compared to a regular clinical examination. MRI is used as the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older, presenting with shoulder pain, and seen in the Duke Sports Medicine clinic by Dr. Wittstein or Dr. Lassiter

Exclusion Criteria:

* Patient cannot have had prior shoulder arthroplasty, instability or history of fracture/dislocation. Pregnant women will be excluded from the study because there will be an MRI. Anyone unable or unwilling to have an MRI will be excluded from the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 40 with shoulder pain that can be MRIed
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Agreement with MRI findings as they pertain to presence or absence of a rotator cuff tear | Within 1 month of exam
  % of exams that agreed with the MRI findings

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn Wittstein, MD, Principal Investigator — Duke Health
Locations (2):
- United States (2):
  - Southeastern Orthopedics Shoulder Center, Raleigh, North Carolina
  - Duke Health Heritage, Wake Forest, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bradley KE, Cook C, Reinke EK, Vinson EN, Mather RC 3rd, Riboh J, Lassiter T, Wittstein JR. Comparison of the accuracy of telehealth examination versus clinical examination in the detection of shoulder pathology. J Shoulder Elbow Surg. 2021 May;30(5):1042-1052. doi: 10.1016/j.jse.2020.08.016. Epub 2020 Aug 29. PMID 32871264